CLINICAL TRIAL: NCT04628676
Title: Comparison of the Efficacy of Irrigation With Epinephrine or Tranexamic Acid on Visual Clarity During Arthroscopic Rotator Cuff Repair: A Randomized Double-Blind Study
Brief Title: Comparison of the Efficacy of Irrigation With Epinephrine or Tranexamic Acid on Visual Clarity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, erhan bayram, medical doctor, Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: saglik bilimleri university
Record Dates: First submitted 2020-10-29; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Rotator Cuff Tears
Keywords: shoulder arthroscopy; irrigation; epinephrine; image quality; tranexamic acid; cuff tear repair; visual clarity
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA group (Experimental): tranexamic acid added to irrigation solution
  Interventions: Drug: tranexamic acid
- EPN group (Experimental): epinephrine added to irrigation solution
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: tranexamic acid — Tranexamic acid is added to the irrigation fluid used in arthroscopic shoulder surgery.
  Other Names: TRANSAMINE %5 5 ml 250 mg
  Arms: TXA group
Drug: Epinephrine — Epinephrine is added to the irrigation fluid used in arthroscopic shoulder surgery.
  Other Names: ADRENALIN 0,5 mg/1 m
  Arms: EPN group

SUMMARY:
The primary aim of this report is to determine whether there is a difference between Epinephrine and Tranexamic acid in providing visual clarity during arthroscopic rotator cuff tear repair.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years

  * American Society of Anesthesiologist Physical Status Classification System : 1-2
  * Undergoing a full arthroscopic double-row repair due to full-thickness cuff tear
  * Being willing to participate the study

Exclusion Criteria:

* • Age < 18 years

  * American Society of Anesthesiologist Physical Status Classification System ≥3
  * Concomitant cardiac diseases
  * Concomitant bleeding disorder or coagulopathy
  * Diabetes mellitus
  * Being pregnant
  * Use of contraceptive pills
  * A history of previous shoulder surgery
  * Uncontrolled hypertension during the operation (>180/110 mm Hg)
  * Unrepairable rotator cuff tears
  * Being unwilling to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | through study completion, an average of 2 year
  Visual analog scale will be rated by surgeon. While 0 is the worst score with no clear vision, 10 was noted as the best score for visual clarity.

SECONDARY OUTCOMES:
total operating time | through study completion, an average of 2 year
  period in minutes from the time the arthroscope was inserted into the glenohumeral joint until the termination of the arthroscopic procedure
average mean arterial pressure | through study completion, an average of 2 year
  mean arterial pressure per operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)